CLINICAL TRIAL: NCT05941260
Title: Standardization of Prostatic Resection Operative Techniques by Virtual Computational Reconstruction and Computational Flow Dynamics
Brief Title: Standardization of Prostatic Resection by Virtual Computational Reconstruction and Computational Flow Dynamics
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, principle investigator, Ain Shams University
Other Study IDs: R1131/2023
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Prostate Hyperplasia; Prostatic Diseases; Voiding Disorders
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male patients above the age of 50: All male patients aged 50 or more with benign prostatic hyperplasia who are scheduled for any planned endourological procedure will be included in our study.
  * Routine cystourethroscopy is a standard procedure in any endourological procedure, whatever the type of procedure.
  * With advanced imaging technology, it is possible through 3D scanning processes of analyzing photos and videos and digitally defining depth, to create 3D models of the tissues and channels, from endoscopy videos.
  * We are going to record this diagnostic cysto-urethroscopy of all patients, and we will send these videos for pre-processing and analysis by virtual computational reconstruction, so that an accurate model could be constructed with a digital model of the urethra geometry and a numerical model of the flow inside the urethra.
  Interventions: Diagnostic Test: Computational fluid dynamics (CFD)

INTERVENTIONS:
Diagnostic Test: Computational fluid dynamics (CFD) — - Video recording starts in an antegrade manner starting from the bladder neck through the prostatic urethra and ends after the verumontanum at the external sphincter. Videos were taken with a very slow movement of the endoscope to ensure the sharpness of the data and to prevent complications in post-processing.
  The focal length and zoom of the endoscope camera were set at the beginning and maintained throughout the capturing, while the angle of the lens changes to capture the widest field possible for each targeted area.
  * Computational fluid dynamics (CFD) can then be used to numerically model the behavior of the flow inside the urethra by solving the governing equations of the flow using the finite volume method.
  * Through which we can develop a urodynamic computer model to simulate the bladder-urethral passage and predict the success of the resection undertaken by the surgeon. No extra intervention will be provided to our patients apart from their routine surgery.

SUMMARY:
The enlargement of the prostate is responsible for voiding dysfunction in men, and especially elderly men. The primary surgical treatment for symptomatic benign prostatic hypertrophy (BPH) was transurethral resection of the prostate (TURP).

However, current resection techniques are predominantly experience-based and judgment-based, with little evidence to support the most effective portion of the prostate to be respected. So, the investigators plan through the study to construct a flow diagram to evaluate the amount of tissue needed to be resected to improve voiding flow dynamics.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is an enlargement of the prostate gland that develops in men and is a common cause of voiding dysfunction in elderly patients. It is a major public health concern, causing high morbidity and substantial worsening of men's quality of life. (QOL)

Transurethral resection of the prostate (TURP) is the standard surgical therapy for obstructive prostatic hypertrophy. Various techniques have been suggested for the systematic removal of the adenomatous tissue, all based on the principle that the resection should be done stepwise as bleeding is the surgeon's major problem, leading to loss of visual field and disorientation, it is imperative that resection and hemostasis should both be completed in one area of the prostatic fossa before the next area is tackled. With the development of new techniques for prostate resection that decreases perioperative morbidity, larger sizes of the prostate are being resected, and a new category of patients is considered eligible for such an intervention with a large prostate size of more than 80 gm. However, current resection techniques are predominantly experience-based and judgment-based, with little evidence to support the most effective portion of the prostate to be resected to give us the best voiding outcome postoperative. So, the investigators plan through this study to construct a flow diagram to evaluate the amount of tissue needed to be resected to improve voiding flow dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Age: above 50 years old, undergoing an elective endo-urological procedure

Exclusion Criteria:

1. Neurogenic bladder
2. Previous prostate or urethral surgery
3. Associated urethral stricture

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all male patients aged above 50 with enlarged prostate who will undergo endoscopic surgical intervention for any urological disease will be included in our study.
Study Population: all male patients above the age of 50 years old with an enlarged prostate and undergoing any endourological procedure with perform cystoscopy during the standard endoscopic procedure.
  Routine cystourethroscopy is a standard procedure in any endourological procedure, whatever the type of procedure.
  With advanced imaging technology, it is possible through 3D scanning processes of analyzing photos and videos then digitally defining the depth, to create 3D models of the tissues and channels, from endoscopy videos.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
computerized urodynamic module of the male urethra | 1 month from the time of video recording during surgery.
  Is to formulate a computerized urodynamic module to simulate the bladder-urethral passage, evaluate urine flow, and predict the amount of needed tissue to be resected to improve patient voiding by a computerized module.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher, Cairo, Egypt